CLINICAL TRIAL: NCT00405275
Title: CSP #551 - Rheumatoid Arthritis: Comparison of Active Therapies in Patients With Active Disease Despite Methotrexate Therapy
Brief Title: Rheumatoid Arthritis: Comparison of Active Therapies in Patients With Active Disease Despite Methotrexate Therapy
Acronym: RACAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Rheumatoid Arthritis Investigational Network (RAIN) (Unknown); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 551; Y1-AR-0048-01 (Other: Inter Agency Agreement between NIAMS and DVA)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Rheumatoid Arthritis
Keywords: antineoplastic; antiparasitics; antirheumatics; chronic diseases; clinical trial; connective tissue; double-blind; drug treatment; gastric medications; joint; multi-site trial; musculoskeletal; randomized; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Chronic Disease | interventions — Etanercept; Methotrexate; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Etanercept and Methotrexate. Participants also received placebo hydroxychloroquine and sulfasalazine
  Interventions: Drug: Etanercept; Drug: methotrexate; Drug: Placebo, triple
- Arm 2 (Active Comparator): Hydroxychloroquine, sulfasalazine and methotrexate. Participants also received placebo etanercept.
  Interventions: Drug: methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine; Drug: Placebo, etanercept

INTERVENTIONS:
Drug: Etanercept — etanercept, subcutaneous injection
  Other Names: Enbrel
  Arms: Arm 1
Drug: methotrexate — baseline methotrexate is maintained throughout the study and is not provided by the sponsor
Drug: Sulfasalazine — sulfasalazine, oral
  Arms: Arm 2
Drug: Hydroxychloroquine — hydroxychloroquine, oral
  Other Names: Plaquenil
  Arms: Arm 2
Drug: Placebo, triple — Participants in Etanercept arm (Arm 1) were given placebo hydroxychloroquine and sulfasalazine pills.
  Arms: Arm 1
Drug: Placebo, etanercept — Participants in triple arm (Arm 2) were given placebo etanercept injections.
  Arms: Arm 2

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease of the joints leading to joint destruction, with significant long-term morbidity and mortality. Early treatment of RA patients with disease-modifying antirheumatic drugs (DMARDs) significantly decreases these complications. Methotrexate (MTX) is an excellent, economical first-line DMARD used to treat a majority of RA patients. While most patients respond well to MTX, many continue to have active disease. Therefore, understanding how to best treat RA patients with active disease despite MTX therapy is critically important. Although a number of therapies with significantly different economic implications have been shown to be effective when added to MTX, no trial has directly compared active therapies. This study will compare therapeutic strategies using two regimens with proven efficacy when added to MTX therapy; a) hydroxychloroquine and sulfasalazine (cost ~ $1000 per year); b) the tumor necrosis factor inhibitor, etanercept (cost ~ $12,000 per year).

We propose a bi-national multi-center randomized, double-blind equivalency trial comparing (A) the strategy of initially adding hydroxychloroquine and sulfasalazine to MTX in patients with active disease despite MTX, with a switch at 24 weeks to etanercept in nonresponders to (B) a strategy of adding etanercept to MTX, with a switch to hydroxychloroquine and sulfasalazine in nonresponders at 24 weeks. If we find that the strategy of first adding hydroxychloroquine and sulfasalazine to MTX identifies a subset of responsive patients and that there is no harm to nonresponders because of early rescue with etanercept, then this less expensive option should become the standard treatment for MTX resistant patients.

Four hundred and fifty RA patients with active disease despite treatment with MTX as indicated by a Disease Activity Score with 28 joints (DAS28) of >4.4 units will be randomized. A DAS improvement of <1.2 (validated as clinically significant) at 24 weeks will be used to identify early nonresponder who will switch therapy. Subjects with a DAS28 improvement of > 1.2 at 24 weeks will remain on their initial therapy. The primary endpoint is the change of DAS 28 scores from baseline to 48 weeks. The secondary endpoint is comparison of radiographic progression of disease at 48 weeks, as measured by the change in Sharp score. Economic and functional outcomes will be assessed and a serum and DNA bank will be established to evaluate potential biomarkers predictive of treatment response/toxicity and disease progression. This trial will recruit 450 subjects over 40 months. At the end of the 48 week blinded active therapy portion of the trial, the blind will be broken and data will be collected in an open fashion until all 450 patients have completed the 48 week portion of the trial.

DETAILED DESCRIPTION:
The main objective of this proposal is to compare two successful treatment strategies that have significantly different economic implications head-to-head in patients with rheumatoid arthritis who have active disease despite methotrexate therapy.

Rheumatoid arthritis (RA) is a chronic inflammatory disease of the joints leading to joint destruction, with significant long-term morbidity and mortality. Early treatment of RA patients with disease-modifying antirheumatic drugs (DMARDs) significantly decreases these complications. Methotrexate (MTX) is an excellent, economical first-line DMARD used to treat a majority of RA patients. While most patients respond well to MTX, many continue to have active disease. Therefore, understanding how to best treat RA patients with active disease despite MTX therapy is critically important. Although a number of therapies with significantly different economic implications have been shown to be effective when added to MTX, no trial has directly compared active therapies. This study will compare therapeutic strategies using two regimens with proven efficacy when added to MTX therapy; a) hydroxychloroquine and sulfasalazine (cost ~ $1000 per year); b) the tumor necrosis factor inhibitor, etanercept (cost ~ $12,000 per year).

We propose a bi-national multi-center randomized, double-blind equivalency trial comparing (A) the strategy of initially adding hydroxychloroquine and sulfasalazine to MTX in patients with active disease despite MTX, with a switch at 24 weeks to etanercept in nonresponders to (B) a strategy of adding etanercept to MTX, with a switch to hydroxychloroquine and sulfasalazine in nonresponders at 24 weeks. If we find that the strategy of first adding hydroxychloroquine and sulfasalazine to MTX identifies a subset of responsive patients and that there is no harm to nonresponders because of early rescue with etanercept, then this less expensive option should become the standard treatment for MTX resistant patients.

Four hundred and fifty RA patients with active disease despite treatment with MTX as indicated by a Disease Activity Score with 28 joints (DAS28) of greater than or equal to 4.4 units will be randomized. A DAS improvement of greater than or equal to 1.2 (validated as clinically significant) at 24 weeks will be used to identify early nonresponder who will switch therapy. Subjects with a DAS28 improvement of ≥ 1.2 at 24 weeks will remain on their initial therapy. The primary endpoint is the change of DAS 28 scores from baseline to 48 weeks. The secondary endpoint is comparison of radiographic progression of disease at 48 weeks, as measured by the change in Sharp score. Economic and functional outcomes will be assessed and a serum and DNA bank will be established to evaluate potential biomarkers predictive of treatment response/toxicity and disease progression. This trial will recruit 450 subjects over 40 months. At the end of the 48 week blinded active therapy portion of the trial, the blind will be broken and data will be collected in an open fashion until all 450 patients have completed the 48 week portion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients must fulfill ACR classification criteria for rheumatoid arthritis.
* All patients must have been 16 years of age or older at time of diagnosis of rheumatoid arthritis.
* All patients must be 18 years of age or older at the time of entry into the study.
* All patients will have been receiving oral or subcutaneous methotrexate 15 to 25 mg/week (unless intolerant and on a minimum 10 mg/week) at a constant dose for at least 4 weeks, and on any methotrexate for no less than 12 weeks.
* All patients will have active disease as defined by a DAS28 of greater than or equal to 4.4.
* If patients are receiving corticosteroids, they must have been on stable dose (less than or equal to 10 mg prednisone or equivalent) for at least two weeks prior to screening.
* If patients are using non-steroidal anti-inflammatory drugs (NSAIDs), they must be on stable doses for at least one week prior to screening.
* If patients have taken leflunomide, cyclosporine, gold, Anakinra, azathioprine, or penicillamine in combination with methotrexate, they must have stopped this therapy at least 8 weeks prior to randomization.
* Laboratory tests must meet the following criteria within 2 weeks of randomization:

  * Serum creatinine 1.8 mg/dL
  * Hemoglobin 9 g/dL
  * WBC 3000 mc/L
  * Neutrophils 1000 mc/L
  * Platelets 100,000 mc/L
  * Serum transaminase level (AST or ALT, whichever is followed at the site) not exceeding 1.2 times upper limit of normal.
  * Albumin no less than 1.0 g/dL (10 g/L) below lower limit of normal. Anything below lower limit of normal must have been stable (or improving) for no less than 90 days. Stable is defined as changes of no more than 0.2 g/dL (2 g/L).
* All patients must be capable of giving informed consent and able to adhere to study visit schedule.
* Subject or designee must have the ability to self-inject investigational product or have a caregiver who can inject subcutaneous injections
* Subjects must meet one of the following criteria with regard to tuberculosis. PPD must be within 180 days of randomization if the patient has no recent exposure/travel history, or within 90 days if the patient has a recent exposure/travel history.

  * Negative PPD; or
  * Positive PPD <5 mm, with a negative chest x-ray; or
  * Positive PPD >5mm, treated for at least 28 days with INH.
* Subjects with an Erythrocyte sedimentation rate (ESR) of less than or equal to 10 and a tender and swollen joint count of at least 10 and does not qualify for the study using the DAS28, will be allowed to use the DAS28-CRP rather than the traditional DAS28 to determine eligibility.

Exclusion Criteria:

* Previous intolerance to methotrexate (unless able to tolerate at least 10 mg/week)
* Sensitivity to study medications
* Previous treatment with methotrexate, sulfasalazine or hydroxychloroquine in combination with each other for longer than 4 weeks duration. No combination use is allowed within 4 weeks of screening.
* No bed or wheelchair-bound patients
* Previous treatment with a TNF- inhibitor (etanercept, infliximab or adalimumab) for more than 5 weeks of therapy. Previous treatment with TNF- inhibitor must have been stopped for reasons other than toxicity or efficacy. No TNF- inhibitor therapy is allowed within the following time frames:

  * Last dose of etanercept must have been at least 4 weeks before screening.
  * Last dose of adalimumab or infliximab must have been at least 8 weeks prior to screening.

Example of an eligible patient: A patient found he could not afford the co-pays for a TNF inhibitor after two doses and stopped taking the medication two months before being evaluated for this trial.

* Evidence of important acute or chronic infections (no IV antibiotics within 1 month, and no PO antibiotics within 2 weeks)
* Pregnant or nursing women
* Women of childbearing potential or their partners who are not practicing an acceptable form of birth control as defined by investigator
* Active substance abuse or psychiatric illness likely to interfere with protocol completion
* History of multiple sclerosis, transverse myelitis, or optic neuritis
* History of macular degeneration unless patient has letter from their ophthalmologist that will allow for participation in trial
* New York Heart Association Class III or IV congestive heart failure
* Active malignancy (other than in situ cervical cancer or non-melanoma skin cancer), or history of lymphoma
* History of HIV
* History of any opportunistic infection - to include but not limited to Pneumocystis carinii, aspergillosis, histoplasmosis, or atypical mycobacterium
* History of porphyria
* Diagnosis of SLE or seronegative spondyloarthropathy or any other form of concomitant arthritis (osteoarthritis is permitted)
* Diagnosis of psoriasis unless rheumatoid factor positive
* Any significant unstable medical condition considered a contraindication by investigator
* Any participation in another investigational drug study during the 90 days preceding randomization.
* Receipt of a live vaccine within 90 days of study entry.
* History of oral or IV cyclophosphamide use
* Life expectancy less than 2 years
* Receipt of steroid injection, intravenous, intramuscular, or intraarticular, within 30 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. O'Dell, Study Chair — VA Medical Center, Omaha
Locations (37):
- United States (28):
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Medical Center, San Francisco, San Francisco, California
  - Pacific Arthritis Center (RAIN), Santa Maria, California
  - VA Greater Los Angeles HCS, Sepulveda, Sepulveda, California
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - St. Mary's/ Duluth Clinic Health System (RAIN), Duluth, Minnesota
  - Park Nicollet (RAIN), Minneapolis, Minnesota
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - VA Medical Center, St Louis, St Louis, Missouri
  - Lincoln Medical Center, Lincoln, Nebraska
  - VA Medical Center, Omaha, Omaha, Nebraska
  - Univesity of Nebraska Medical Center, Omaha, Nebraska
  - Bone, Spine Sports Clinic (RAIN), Bismarck, North Dakota
  - VA Medical Center, Fargo, Fargo, North Dakota
  - VA Medical Center, Portland, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - State College, State College, Pennsylvania
  - Geisinger Medical Group- Wilkes Barre, Wyoming Valley, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - Rapid City Medical Center (RAIN), Rapid City, South Dakota
  - Avera Research Institute (RAIN), Sioux Falls, South Dakota
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Medical & Regional Office Center, White River, White River Junction, Vermont
- Canada (9):
  - University of Calgary (CRRC), Calgary, Alberta
  - University of Manitoba (CRRC), Winnipeg, Manitoba
  - Brampton (CRRC), Brampton, Ontario
  - Credit Valley Rheumatology, Missassauga, Ontario
  - Newmarket (CRRC), Newmarket, Ontario
  - Mount Sinai Hospital (CRRC), Toronto, Ontario
  - Clinical Research and Arthritis Center, Windsor, Ontario
  - Hopital Notre Dame (CRRC), Montreal, Quebec
  - Crc-Chus (Crrc), Sherbrooke, Quebec

REFERENCES:
- [Result] O'Dell JR, Mikuls TR, Taylor TH, Ahluwalia V, Brophy M, Warren SR, Lew RA, Cannella AC, Kunkel G, Phibbs CS, Anis AH, Leatherman S, Keystone E; CSP 551 RACAT Investigators. Therapies for active rheumatoid arthritis after methotrexate failure. N Engl J Med. 2013 Jul 25;369(4):307-18. doi: 10.1056/NEJMoa1303006. Epub 2013 Jun 11. PMID 23755969
- [Derived] Peper SM, Lew R, Mikuls T, Brophy M, Rybin D, Wu H, O'Dell J. Rheumatoid Arthritis Treatment After Methotrexate: The Durability of Triple Therapy Versus Etanercept. Arthritis Care Res (Hoboken). 2017 Oct;69(10):1467-1472. doi: 10.1002/acr.23255. Epub 2017 Sep 6. PMID 28388820
- [Derived] Quach LT, Chang BH, Brophy MT, Soe Thwin S, Hannagan K, O'Dell JR. Rheumatoid arthritis triple therapy compared with etanercept: difference in infectious and gastrointestinal adverse events. Rheumatology (Oxford). 2017 Mar 1;56(3):378-383. doi: 10.1093/rheumatology/kew412. PMID 27994091
- [Derived] Bansback N, Keystone E, O'Dell J, Phibbs CS, Hannagan K, Brophy M, Anis A. Making smart investment decisions in clinical research. Trials. 2015 Dec 29;16:590. doi: 10.1186/s13063-015-1123-1. PMID 26712327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bi-national, multi-center 3.5 year recruitment at 16 VA, 12 RAIN and 8 Canadian medical centers.
Groups:
- Triple: Hydroxychloroquine (400mg daily); Sulfasalazine (1g daily for 6 weeks, then increased to 2g daily; Methotrexate (maintaining baseline dose, 10-25mg weekly); Placebo, etanercept (subcutaneous injection).
  Nonresponders (change in DAS28 < 1.2units at 24 weeks) were switched to Etanercept at 24 weeks. This is denoted in results table below as "switch". "No switch" participants remained on Triple therapy throughout the trial.
- Etanercept: Etanercept (50mg subcutaneous injections weekly); Methotrexate (maintaining baseline dose, 10-25mg weekly); Placebo, triple: placebo hydroxychloroquine (tablets daily) and placebo sulfasalazine (tablets daily).
  Nonresponders (change in DAS28 < 1.2units at 24 weeks) were switched to Triple. This is denoted in results table below as "switch". "No switch" participants remained on Etanercept therapy throughout the trial.
Period: Overall Study
Arm/Group | Triple | Etanercept
Started | 178 | 175
24 Weeks (Total) | 163 | 165
24 Week (no Switch) | 119 | 121
24 Week (Switch) | 44 | 44
Completed | 155 | 156
Not Completed | 23 | 19
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Unwilling to continue | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Triple: Hydroxychloroquine, sulfasalazine and methotrexate
- Etanercept: Etanercept and Methotrexate
- Total: Total of all reporting groups
Arm/Group | Triple | Etanercept | Total
Number analyzed (Participants) | 178 | 175 | 353
Age Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.0) | 56.0 (13.2) | 56.9 (13.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 77 | 85 | 162
  Male | 101 | 89 | 190
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 134 | 130 | 264
  Canada | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Mean 48-week Change in DAS28
Description: Average difference between 48-week and Baseline DAS28.
  The Disease Activity Score for 28 Joints (DAS28) is a well-validated composite outcome measure ranging from 2-10 (higher scores indicating more disease) that incorporates a tender and swollen joint count of 28 joints, a laboratory measure of systemic inflammation (ESR) and a patient-reported general assessment of health on a visual analog scale (ranging from 0-10cm) all into one measure.
  Low disease activity is defined as DAS28 ≤ 3.2 units.
Time Frame: 48 weeks after baseline assessment
Population: Intention to treat analysis was performed on participants with Week 48 DAS28 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triple | Etanercept
Number analyzed (Participants) | 154 | 155
units on a scale | -2.12 (1.28) | -2.29 (1.30)

ADVERSE EVENTS:
Time Frame: Beginning at Informed Consent until each participant's last study follow-up contact (expected to be 48 weeks), including a period of 30 days after last contact for SAE reporting.
Description: Serious and non-serious Adverse Events are reported according to treatment at the time of event. Participants that switched therapies are represented in both treatments. Participants were seen every 6 weeks for adverse event monitoring.
Arm/Group | Triple | Etanercept
Serious Adverse Events (participants affected / at risk) | 38/222 | 43/219
Other Adverse Events (participants affected / at risk) | 40/222 | 55/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple (N=222) | Etanercept (N=219)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6) | 7 (7)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Catheterisation cardiac normal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Treatment noncompliance (Social circumstances) | 0 (0) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple (N=222) | Etanercept (N=219)
Nausea (Gastrointestinal disorders) | 16 (23) | 17 (18)
Nasopharyngitis (Infections and infestations) | 8 (8) | 14 (16)
Upper respiratory tract infection (Infections and infestations) | 12 (17) | 19 (23)
Headache (Nervous system disorders) | 17 (20) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dr. O'Dell is an employee of the Sponsor. Dr. Edward Keystone is not.

Per the signed Investigator Agreement, PIs agreed to "maintaining the confidentiality of study data and not publishing study data without prior approval of the study's Executive Committee".